CLINICAL TRIAL: NCT01461915
Title: A Randomized Phase II Open Label Study to Assess the Efficacy & Safety of Gemcitabine + Abraxane® With or Without ODSH (2-0, 3-0 Desulfated Heparin) as First Line Treatment of Metastatic Pancreatic Cancer
Brief Title: Phase 2 Study to Assess the Efficacy & Safety of Gemcitabine + Nab Paclitaxel With or Without Dociparstat in Metastatic Pancreatic Cancer Patients
Acronym: PGPC1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Collaborators: Translational Drug Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PGX-ODSH-2011-PC1
Record Dates: First submitted 2011-10-13; First posted 2011-10-28 (Estimated); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Taxes; Albumin-Bound Paclitaxel; Gemcitabine; N-desulfated,2-O,3-O-desulfated heparin

ARMS (3):
- Run-in (Experimental): During the Run-In Period, patients will receive gemcitabine + nab-paclitaxel + dociparstat to assess the compatibility of the combination.
  • Nab-paclitaxel + gemcitabine + dociparstat:
  * Nab-paclitaxel 125 mg/m2 will be administered intravenously (IV) over 30 minutes followed by the administration of gemcitabine IV infusion at 1000 mg/m2 over 30 minutes. Nab paclitaxel + gemcitabine will be administered weekly for 3 weeks followed by 1 week of rest (28-day cycle).
  * Dociparstat IV bolus at 4 mg/kg will be administered in 5 minutes immediately following the completion of gemcitabine administration.
  * Dociparstat 48-hour IV continuous infusion at 0.375 mg/kg/hr will be administered immediately following the dociparstat IV bolus administration.
  Interventions: Drug: Nab paclitaxel; Drug: Gemcitabine; Drug: Dociparstat
- Arm A (Experimental): Patients randomized to Arm A will receive gemcitabine + nab-paclitaxel + dociparstat.
  • Nab-paclitaxel + gemcitabine + dociparstat:
  * Nab-paclitaxel 125 mg/m2 will be administered IV over 30 minutes followed by the administration of gemcitabine IV infusion at 1000 mg/m2 over 30 minutes. Nab paclitaxel + gemcitabine will be administered weekly for 3 weeks followed by 1 week of rest (28-day cycle).
  * Dociparstat IV bolus at 4 mg/kg will be administered in 5 minutes immediately following the completion of gemcitabine administration.
  * Dociparstat 48-hour IV continuous infusion at 0.375 mg/kg/hr will be administered immediately following the dociparstat IV bolus administration.
  Interventions: Drug: Nab paclitaxel; Drug: Gemcitabine; Drug: Dociparstat
- Arm B (Active Comparator): Patients randomized to Arm B will receive gemcitabine + nab-paclitaxel. • Nab-paclitaxel + gemcitabine:
  o Nab-paclitaxel 125 mg/m2 will be administered IV over 30 minutes followed by the administration of gemcitabine IV infusion at 1000 mg/m2 over 30 minutes. Nab paclitaxel + gemcitabine will be administered weekly for 3 weeks followed by 1 week of rest (28-day cycle).
  Interventions: Drug: Nab paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: Nab paclitaxel — Nab-paclitaxel 125 mg/m2 will be administered IV over 30 minutes. Nab-paclitaxel will be administered weekly for 3 weeks followed by 1 week of rest (28-day cycle).
  Other Names: Abraxane
Drug: Gemcitabine — Following the completion of nab-paclitaxel administration, gemcitabine IV infusion at 1000 mg/m2 will be administered over 30 minutes. Gemcitabine will be administered weekly for 3 weeks followed by 1 week of rest (28-cycle).
Drug: Dociparstat — Following the completion of gemcitabine administration, dociparstat IV bolus at 4 mg/kg will be administered in 5 minutes immediately after completion of gemcitabine administration. Immediately following the dociparstat IV bolus administration, dociparstat 48-hour IV continuous infusion at 0.375 mg/kg/hr will be administered.
  Other Names: ODSH; 2-O, 3-O Desulfated Heparin; Dociparstat sodium
  Arms: Arm A; Run-in

SUMMARY:
This randomized, Phase 2, open label study aims to assess the efficacy and safety of gemcitabine + nab paclitaxel with or without dociparstat (ODSH) as first line treatment of metastatic pancreatic cancer. This study consists of 2 periods: a Run-in Period and a Randomized Period.

DETAILED DESCRIPTION:
Dociparstat (ODSH) has demonstrated in vitro and in vivo inhibitory activity on mechanisms that are believed to play important roles in pancreatic cancer invasion, metastasis, and resistance to chemotherapy and radiation. Pancreatic cancer appears to have a dependence on autophagy, a regulated catabolic pathway to degrade and recycle cellular organelles and macromolecules. Autophagy appears to be largely driven by the binding of high mobility group box-1 protein (HMGB1) to the receptor for advanced glycation end-products (RAGE), which is strongly inhibited by dociparstat. Autophagy appears to not only assist pancreatic cancer cells to survive in a hypoxic, relatively avascular environment, but also appears to play an important role in chemotherapy resistance. Other important biological activities promoting pancreatic cancer invasion and metastasis affected by dociparstat include the inhibition of heparanase and the binding of tumor cells to endothelium and platelets mediated by the selectins. It is believed that these biological activities such as the inhibition of RAGE, heparanase, and selectin-mediated metastasis, can be inhibited by dociparstat at dose levels that can safely be administered without clinically significant anticoagulation.

The standard of care of pancreatic cancer is evolving. It appears that 2 combination regimens, the "FOLFIRINOX" regimen (a combination of 5-fluorouracil, leucovorin, irinotecan and oxaliplatin) and the combination of gemcitabine + nab-paclitaxel, could have more activity than the previous standard treatment of gemcitabine alone.

Patients with advanced metastatic pancreatic cancer who have not received chemotherapy, surgical or radiation treatments and have a good performance status are eligible to participate in this study. This study consists of 2 periods: a Run-in Period and a Randomized Period. In total, 10 patients are planned to be enrolled in a Run-in Period to receive gemcitabine + nab-paclitaxel + dociparstat. Pharmacokinetic sampling and safety assessments are to be conducted to decide on the continuation to the Randomized Period of the study where 50 patients are planned to be randomized at a 1:1 ratio to either of the 2 study arms:

* Arm A: Patients will receive gemcitabine + nab-paclitaxel + dociparstat
* Arm B: Patients will receive gemcitabine + nab-paclitaxel

The primary endpoint of this study is mean progression free survival. The secondary endpoints of this study are to consist of tumor response by Response Evaluation Criteria in Solid Tumors (RECIST) criteria, overall survival at the end of the study, and changes from baseline for carbohydrate antigen (CA) 19-9 marker, weight, and plasma albumin.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all the following criteria to be eligible for this study:

1. Has histologically confirmed adenocarcinoma of the pancreas that is metastatic and for which potential curative measures, such as resection of an isolated metastasis, are not available. Patients with islet cell neoplasms will be excluded.
2. Has ≥ 1 metastatic tumors measurable by computerized tomography (CT) scan AND a serum carbohydrate antigen (CA) 19-9 measurement >2 times the upper limit of normal. Patients must have measurable disease, defined as at least 1 lesion that could be accurately measured in at least 1 dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >20 mm with conventional techniques or as >10 mm with spiral CT scan.
3. Is male or non-pregnant and non-lactating female and ≥ 18 to ≤ 75 years of age. If a female patient is of child-bearing potential, she must have a negative serum pregnancy test documented within 72 hours prior to the first administration of study drug and on Day 1 of each cycle thereafter. If sexually active, the patient must agree to use contraception prior to study entry and for the duration of study participation.
4. Must have received no prior radiotherapy or chemotherapy for metastatic disease. Patients who have received radiotherapy or chemotherapy as adjuvant or neo-adjuvant therapy for locally advanced disease 6 months or more prior to enrollment into this study are eligible.
5. Has adequate biological parameters as demonstrated by the following blood counts at Screening (obtained ≤14 days prior to randomization) and at Baseline-Day 0: Absolute neutrophil count (ANC) ≥1.5 × 109/L; Platelet count ≥ 100,000/mm3 (100 × 109/L); Hemoglobin (Hgb) ≥ 9 g/dL.
6. Has the following blood chemistry levels at Screening (obtained ≤14 days prior to randomization) and at Baseline-Day 0:

   * Aspartate aminotransferase (AST; SGOT), alanine aminotransferase (ALT; SGPT) ≤ 2.5 × upper limit of normal range (ULN), unless liver metastases are present, then ≤5 × ULN is allowed. Total bilirubin ≤1.5 × ULN.
   * Serum creatinine (Cr) within normal limits or calculated clearance ≥60 mL/min/1.73 m2 for patients with creatinine (Cr) levels above or below the institutional normal value. If using Cr clearance, actual body weight should be used for calculating Cr clearance (e.g., using the Cockcroft-Gault formula).
7. Has acceptable coagulation studies at Screening (obtained ≤14 days prior to randomization) as demonstrated by prothrombin time (PT) and partial thromboplastin time (PTT) within normal limits (±15%).
8. Has an Eastern Cooperative Oncology Group (ECOG) performance status score of ≤1.
9. Has been informed about the nature of the study, and agrees to participate in the study, and signed the Informed Consent Form (ICF) prior to participation in any study-related activities.

Exclusion Criteria:

If a patient meets any of the following criteria, they are not eligible to participate in this study:

1. Has brain metastases.
2. Has only locally advanced disease.
3. Has experienced an increase of ECOG score to >1 between Screening and Randomization.
4. Requires continuous treatment with coumadin or other oral or parenteral anticoagulation (heparin, low molecular weight heparin [LMWH], heparinoids) to prevent or treat thromboembolic disease. The use of prophylactic antiplatelet drugs such as clopidogrel and aspirin are allowed before and during the study.
5. Has active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy.
6. Has undergone major surgery, other than diagnostic surgery (i.e., surgery done to obtain a biopsy for diagnosis without removal of an organ), within 4 weeks prior to Randomization in this study.
7. Has a history of allergy or hypersensitivity to any of the study drugs, their pharmaceutical class, or any of their excipients.
8. Has a concomitant serious medical or psychiatric illness that, in the opinion of the Investigator, could compromise the patient's safety or the study data integrity.
9. Is enrolled in any other clinical protocol or investigational trial that involves administration of anti-neoplastic compounds for the treatment of metastatic pancreatic cancer.
10. Is unwilling or unable to comply with study procedures.
11. Nab-paclitaxel is metabolized by cytochrome P450 (CYP) 2C8 and CYP3A4. Co-administration of substrates, inhibitors of CYP2C8 and/or CYP3A4 with nab-paclitaxel is not allowed. The following medications and substances are not allowed during the study: ritonavir, saquinavir, indinavir, nelfinavir, rifampicin, carbamazepine, phenytoin, efavirenz, or nevirapine, grapefruit (juice or seeds) or some herbals like St. John's wort.
12. Has risk factors for or a history of Torsades des Pointes (TdP), or a significant QT prolongation that, in the opinion of the Investigator, may place the patient at risk.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-11; Primary Completion 2012-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Number of Patients who Achieved Progression-Free Survival | 9 months
  The primary objective of this study is to evaluate progression-free survival (PFS) according to Response Evaluation Criteria In Solid Tumors (RECIST) Guidelines Version 1.1. This will be assessed from Baseline to disease progression or death (whichever occurred first), for up to 9 months.

SECONDARY OUTCOMES:
Proportion of Patients who Achieved Overall Survival | 9 months
  A secondary objective of this study is to evaluate overall survival at the End of the Study.

CONTACTS AND LOCATIONS:
Overall Officials: Mitesh J Borad, MD, Principal Investigator — Division of Hematology/Oncology, Department of Internal Medicine, Mayo Clinic , Scottsdale Arizona; Stephen Marcus, MD, Study Director — ParinGenix Inc, Weston FL
Locations (16):
- United States (16):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Disney Family Cancer Center, Burbank, California
  - Marin Cancer Care, Greenbrae, California
  - Scripps Clinic Torrey Pines ( Green Hospital), La Jolla, California
  - Cleveland Clinic Florida, Weston, Florida
  - Loyola University Medical Center/Cardinal Bernardin Cancer Center, Maywood, Illinois
  - Indiana University Health, Goshen Center for Cancer Care, Goshen, Indiana
  - Fesit-Weiller Cancer Center, Shreveport, Louisiana
  - Saint Mary's Health Care, Grand Rapids, Michigan
  - Summa Health System - Cooper Cancer Center, Akron, Ohio
  - Thomas Jefferson University [Kimmel Cancer Center], Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UPMC Cancer Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina Hollings Cancer Center, Charleston, South Carolina
  - University of Texas Medical Branch, Galveston, Texas
  - South Texas Oncology & Hematology, San Antonio, Texas

REFERENCES:
- [Background] Von Hoff DD, Ramanathan RK, Borad MJ, Laheru DA, Smith LS, Wood TE, Korn RL, Desai N, Trieu V, Iglesias JL, Zhang H, Soon-Shiong P, Shi T, Rajeshkumar NV, Maitra A, Hidalgo M. Gemcitabine plus nab-paclitaxel is an active regimen in patients with advanced pancreatic cancer: a phase I/II trial. J Clin Oncol. 2011 Dec 1;29(34):4548-54. doi: 10.1200/JCO.2011.36.5742. Epub 2011 Oct 3. PMID 21969517